CLINICAL TRIAL: NCT07130955
Title: To Evaluate the Efficacy and Safety of Six-Channel Radiofrequency Ablation System for Renal Denervation in Patients With Uncontrolled Hypertension Combined With Chronic Kidney Disease
Brief Title: A Randomized Trial of Six-Channel RF Ablation System for Renal Denervation in Uncontrolled Hypertension and Chronic Kidney Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Golden Leaf MedTec Co. Ltd (Industry)
Collaborators: Beijing Anzhen Hospital (Other); Shanghai Zhongshan Hospital (Other); Guangdong Provincial People's Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); West China Hospital (Other); Jiangxi Provincial People's Hopital (Other); Navy General Hospital, Beijing (Other); Qilu Hospital of Shandong University (Other); Xijing Hospital (Other); Fujian Provincial Hospital (Other); First Affiliated Hospital of Fujian Medical University (Other); Henan Provincial People's Hospital (Other); Hebei Provincial People's Hospital (Unknown); Anhui Provincial Hospital (Other Government); The First Hospital of Jilin University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Qianfoshan Hospital (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Mianyang Central Hospital (Other); The Third People's Hospital of Chengdu (Other); General Hospital of the Eastern Theater Command (Unknown); China-Japan Union Hospital, Jilin University (Other); Shanxi Bethune Hospital (Other); Second Hospital of Shanxi Medical University (Other); Yan'an Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MLWY-S20250422
Record Dates: First submitted 2025-07-28; First posted 2025-08-19 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-08

CONDITIONS: Hypertension; CKD - Chronic Kidney Disease
Keywords: Uncontrolled Hypertension; CKD; RDN
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Prospective, Multicenter, Randomized, Parallel-Controlled,The trial will enroll 236 subjects (trial group: control group = 1:1).
Who Masked: Participant
Masking Description: The trial will enroll 236 subjects (trial group: control group = 1:1)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Renal Denervation (RDN) (Experimental): Participants receive percutaneous renal sympathetic denervation under digital subtraction angiography (DSA) guidance using a six-channel radiofrequency generator(model 25D1G, software release SRG-V1) and ultra-guiding radiofrequency denervation catheter (model 25C6W127F115T) manufactured by Shanghai Golden Leaf MedTec Co., Ltd(BRATTEA). All participants receive a standardized antihypertensive regimen for ≥4 weeks before the procedure and thereafter per protocol. Follow-up visits occur at 7 days or before discharge, and at 1, 3, 6, 12, 24, and 36 months.
  Assigned Interventions: Device: Six-channel RF Renal Denervation System; Drug: Standardized Antihypertensive Therapy
  Interventions: Device: Six-channel RF Renal Denervation System
- Parallel control with sham operation (Sham Comparator): Participants undergo a sham procedure: femoral artery puncture and selective renal angiography under DSA guidance are performed. The RF generator is connected to a dummy load, and activation sounds are emitted, but no energy is delivered. Participants remain on the procedure table for at least 35 minutes before sheath removal. Background standardized antihypertensive therapy is provided for ≥4 weeks pre-procedure and continued per protocol. Follow-up visits occur at 7 days or before discharge, and at 1, 3, 6, and 12 months. After completing the 6-month visit, participants may transition to active RDN and then be followed up to 36 months; those declining crossover will continue follow-up at 12，24 and 36 months.
  Assigned Interventions: Procedure: Sham operation; Drug: Standardized Antihypertensive Therapy
  Interventions: Procedure: Parallel controln with sham operation(there is no rade and/or generic name,It is a blank control sham operation)

INTERVENTIONS:
Device: Six-channel RF Renal Denervation System — DSA-guided percutaneous renal sympathetic denervation using a six-channel RF renal denervation system-comprising the six-channel radiofrequency generator (specification model: 25D1G, software release version: SRG-V1) and the ultra-guiding radiofrequency denervation catheter (specification model: 25C6W127F115T)
  Arms: Renal Denervation (RDN)
Procedure: Parallel controln with sham operation(there is no rade and/or generic name,It is a blank control sham operation) — Sham procedure including femoral artery puncture and selective renal angiography; the six-channel radiofrequency generator is connected to a dummy load and produces activation sounds, but no energy is delivered. Minimum table time before sheath removal is 35 minutes.
  Arms: Parallel control with sham operation

SUMMARY:
Prospective, Multi-Center, Randomized, Parallel-Controlled, Uptake clinical trial to evaluate the efficacy and safety of the six-channel radiofrequency（RF) renal denervation system-comprising the six-channel radiofrequency generator (specification model: 25D1G, software release version: SRG-V1) and the disposable ultra-guiding radiofrequency denervation catheter (specification model: 25C6W127F115T)-for renal denervation in patients with uncontrolled hypertension and chronic kidney disease.

DETAILED DESCRIPTION:
The six-channel RF renal denervation system, consisting of the six-channel radiofrequency generator (specification model: 25D1G, software release version: SRG-V1) and the disposable ultra-guiding radiofrequency denervation catheter (specification model: 25C6W127F115T), is designed and manufactured by Shanghai Golden Leaf MedTec Co., Ltd (BRATTEA) for renal artery radiofrequency denervation.

This Prospective, Multi-Center, Randomized, parallel-controlled uptake clinical trial aims to evaluate the system's efficacy and safety for renal denervation in patients with uncontrolled hypertension and chronic kidney disease, and to provide clinical evidence supporting the expansion of indications. The trial will be conducted by the Regulations on the Supervision and Administration of Medical Devices, the Measures for the Administration of Medical Device Registration and Filing, the Good Clinical Practice for Medical Devices, and other applicable requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 to 65 years, inclusive, at the time of consent;
2. Hypertensive subjects who have been taking 2 types of standardized antihypertensive drugs continuously and stably for at least 4 weeks, with office systolic blood pressure still ≥150 mmHg and <180 mmHg, and 24-hour ambulatory mean systolic blood pressure (24h SBP) ≥135 mmHg and <170 mmHg; or who have been taking ≥3 types of standardized antihypertensive drugs continuously and stably for at least 4 weeks, with office systolic blood pressure ≥140 mmHg and <180 mmHg, and 24h SBP ≥130 mmHg and <170 mmHg;
3. Estimated glomerular filtration rate (eGFR) ≥20 mL/min/1.73m² and <60 mL/min/1.73m²;
4. The subject or his/her legal representative fully understands the content of the informed consent form for this trial and voluntarily signs the written informed consent form.

Exclusion Criteria:

1. Pregnant or breastfeeding, or planning pregnancy during the study.
2. Renal artery anatomy unsuitable for ablation (e.g., ≥50% stenosis, renal artery aneurysm, malformation, renal artery diameter <3 mm, or treatable segment length <20 mm).
3. Subjects with a solitary kidney, prior renal transplantation, or requiring dialysis.
4. Prior renal artery intervention or prior renal denervation.
5. Other secondary hypertension not related to kidney disease (such as primary aldosteronism, pheochromocytoma/paraganglioma, Cushing's syndrome, thyroid disease, aortic coarctation, monogenic hypertension, renovascular hypertension, etc.).
6. Allergic to contrast agents.
7. Major surgery or trauma within 1 month before enrollment; acute coronary syndrome within 6 months; or planned surgery or cardiovascular interventional therapy within the next 6 months.
8. Orthostatic hypotension.
9. Type 1 diabetes mellitus.
10. Primary pulmonary arterial hypertension.
11. History of bleeding diathesis and haematological disorders or coagulopathy
12. History of thromboembolic event within 6 months.
13. History of stroke or transient ischemic attack (TIA) within 6 months.
14. Severe peripheral arterial disease or unstable abdominal aortic aneurysm.
15. Severe valvular heart disease or anticipated need for surgical valve replacement during the study period.
16. NYHA Class III/IV heart failure at screening or hospitalization for exacerbation of chronic heart failure within the past six months.
17. History of ventricular fibrillation, polymorphic ventricular tachycardia within six months, or prior implantation of an implantable cardioverter-defibrillator (ICD) or pacemaker.
18. Acute kidney injury (AKI) within 4 weeks before enrollment or acute kidney disease ，AKI: ≥50% increase in serum creatinine within 7 days, or absolute increase ≥0.3 mg/dL (≥26.5 μmol/L) within 48 hours, or oliguria (<0.5 mL·kg-¹·h-¹ for ≥6 hours).
19. Severe hepatic dysfunction.
20. Concomitant severe diseases that may interfere with study participation or affect survival, such as malignancy or AIDS.
21. Known drug or alcohol dependence, difficulty understanding the study protocol, inability or unwillingness to comply with follow-up requirements.
22. Current or planned participation in other clinical trials of drugs or medical devices (post-marketing registry studies permitted).
23. Acute or severe systemic infection.
24. Other conditions deemed unsuitable for participation by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in 24-hour Ambulatory Systolic Blood Pressure at Month 6 (ABPM) | Baseline to Month 6 post-procedure
  24-hour mean systolic BP measured by validated ambulatory BP monitoring; change is Month 6 minus Baseline.

SECONDARY OUTCOMES:
Change from Baseline in 24-hour Ambulatory Diastolic Blood Pressure at Month 6 (ABPM) | Baseline to Month 6 post-procedure
  24-hour mean systolic BP measured by validated ambulatory BP monitoring;
Change from Baseline in 24-hour Ambulatory Blood Pressure (including both systolic and diastolic BP) | Baseline to Months 1, 3, 12, 24, and 36 post-procedure
  24-hour mean systolic BP measured by validated ambulatory BP monitoring;
Change from Baseline in Daytime and Nighttime Ambulatory Systolic Blood Pressure (ABPM) | Baseline to Months 1, 3, 6, 12, 24, and 36 post-procedure
  24-hour mean systolic BP measured by validated ambulatory BP monitoring;
Change from Baseline in Office Blood Pressure (including both systolic and diastolic BP) | Baseline to Months 1, 3, 6, 12, 24, and 36 post-procedure
  measured by validated office blood pressure monitoring
Percentage of Participants with 24-hour Ambulatory Systolic BP <130 mmHg | Months 1, 3, 6, 12, 24, and 36 post-procedure
  24-hour mean systolic BP measured by validated ambulatory BP monitoring;
Percentage of subjects with office systolic BP within the target ranges (<140 mmHg and <130 mmHg) | Months 1, 3, 6, 12, 24, and 36 post-procedure
  measured by validated office blood pressure monitoring
Responder Rate: ≥5 mmHg Reduction in 24-hour Ambulatory Systolic BP | Months 1, 3, 6, 12, 24, and 36 post-procedure
  Proportion of participants with a reduction ≥5 mmHg from baseline in 24-hour mean systolic BP by ABPM.
Change from Baseline in Antihypertensive Medication Use | Baseline to hospital discharge or Day 7 (whichever occurs first), and to Months 1, 3, 6, 12, 24, and 36 post-procedure
  Change in the number of concurrently prescribed antihypertensive agents .
Change from Baseline in Cardiac Function (by Echocardiography) | Baseline to Months 1, 3, 6, 12, 24, and 36 post-procedure
  by Echocardiography
Change from Baseline in Heart Rate (by ECG) | Baseline to Months 1, 3, 6, 12, 24, and 36 post-procedure
  Resting heart rate measured by standard 12-lead ECG; change is Follow-up minus Baseline.
Device and Procedure Success | Intra-procedure (Day 0)
  Successful completion of intended renal denervation ablations in eligible segments of the renal arteries without device malfunction requiring replacement or procedure abortion.
Periprocedural major adverse event (MAE) rate | Baseline to 30 days post-procedure
  Hospitalization for a clinically significant hypotensive or hypertensive event;
  Vascular complications requiring surgical repair, endovascular therapy, thrombin injection, or blood transfusion;
  Renal artery dissection or perforation requiring intervention;
  Significant embolic events causing end-organ damage or requiring intervention to prevent it;
  Severe renal impairment (>50% decrease in eGFR or >50% increase in serum creatinine from baseline) or ESRD (eGFR <15 mL/min/1.73 m²);
  All-cause death;
  New renal artery stenosis ≥70% (confirmed by angiography).
Safety event rates | Baseline to Months 36 post-procedure
  Interventional complications: pseudoaneurysm, thrombosis, dissection, AV fistula, rupture or perforation, renal artery stenosis.
  All-cause mortality.
  MACCE: stroke (ischemic or hemorrhagic), ACS (AMI or unstable angina), cardiovascular death.
  Severe renal dysfunction (eGFR decrease >50% or creatinine increase >50% from baseline) or ESRD (eGFR <15 mL/min/1.73 m²).
  New renal artery stenosis ≥70% within 6 months (confirmed by angiography).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No